Cover Page NCT03287635

Clinical Efficacy of H.P. Acthar Gel 80 Units/ml to Improve the Signs and Symptoms in Subjects with Dry Eye Disease

Date May 10, 2018

## Statistical Analysis Plan Acthar Pilot Study

The statistical analysis plan for this study includes analysis of patients completing the trial and measuring the change from baseline to final visit including intervisit changes. For each of these time points, P-values will be collected, standard deviations, standard error means, 95% confidence intervals of the difference and 2-tailed t test applied. There is no placebo or control in this study and the number of participants was not powered to show statistical differences.